CLINICAL TRIAL: NCT00447941
Title: Randomized, Double-blind, Placebo-controlled, Ascending Multiple Dose Study of the Safety, Pharmacokinetics, and Pharmacodynamics of Sca-136 Administered Orally to Healthy Male Japanese Subjects
Brief Title: Safety, PK and PD Study in Healthy Male Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3153A1-103
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: SCA-136

SUMMARY:
Study assessing pharmacokinetics, pharmacodynamics, safety, and tolerability of oral doses of SCA-136 in healthy male Japanese subjects

ELIGIBILITY:
Inclusion Criteria

* Men aged 20 to 45 years at the time of obtaining informed consent.
* Body mass index (BMI) in the range of 18.5 to 25.0 kg/m2 and body weight ≥ 50 kg.
* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG).

Exclusion Criteria

* Presence or history of any disorder that may prevent the successful completion of the study.
* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
* Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion (ADME) of the test article (eg, resection of liver, kidney, or gastrointestinal tract).

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2006-06; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer